CLINICAL TRIAL: NCT04343105
Title: The Effect of Ultrasound-guided Bilateral Single Shot Pecto -Intercostal Plane Block on Recovery After On-pump Coronary Bypass Graft Surgery
Brief Title: Pecto-intercostal Plane Block in On-pump Coronary Bypass Graft Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, tarek abdel hay mostafa, principle investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: pecto-intercostal plane block
Record Dates: First submitted 2020-04-03; First posted 2020-04-13 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Enhanced Recovery After Cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sham group (Sham Comparator): will receive sham bilateral ultrasounded guided single shot pecto-intercostal plane block between 3rd and 4th rib 2 cm lateral to sternal border for each side after induction of anaesthesia in supine position
  Interventions: Procedure: pecto-intercostal plane block
- real group (Experimental): will receive real bilateral ultrasounded guided single shot pecto-intercostal plane block between 3rd and 4th rib 2 cm lateral to sternal border for each side after induction of anaesthesia in supine position with 10 ml bupivacaine 0.5% + 10 ml lidocaine 2% in total volume 20 ml for each side.
  Interventions: Procedure: pecto-intercostal plane block

INTERVENTIONS:
Procedure: pecto-intercostal plane block — under ultrasound guidance, pecto-intercostal plane block will be performed between 3rd and 4th rib 2 cm lateral to sternal border in supine position at the interfascial plane between pectoralis major muscle and intercostal muscles

SUMMARY:
Fast track and ultrafast track cardiac anaesthesia appear to demonstrate improved outcomes without compromising patient safety. Their benefits include shorter intensive care unit stays, reduced duration of mechanical ventilation and lower health care costs. Regional anesthesia has played an important role in enhanced recovery pathways for other surgical services and allows for reduced systemic opioid use during intraoperative and postoperative care This study will be conducted to evaluate the effectiveness and safety of ultrasound guided bilateral single shot pecto - intercostal plane block on recovery after on pump CABG surgery.

DETAILED DESCRIPTION:
Fast-track anesthesia (FTA) is a procedure that enables extubation in intensive care unit (ICU) within 6 h after surgery to facilitate the recovery of consciousness and autonomous breathing. It has been safely applied to cardiac surgery since the 1990s.

FTA is feasible and safe and reduces the occurrence of ventilator induced complications, thereby decreasing ICU stay, resource use and cost.

Ultra-fast tract anesthesia (UFTA) was developed after fast-track anesthesia to further optimize the use of medical resource. With UFTA, extubation is performed immediately or within 1 h after surgery in the operating room. The benefits of UFTA include lower incidence of postoperative complications, better hemodynamic performance, shorter ICU stay.

Fast track and ultrafast track cardiac anaesthesia can be achieved by reduced opioid doses or opioid free with multimodal analgesia augmented with bilateral regional anaesthesia as pecto - intercostal plane block.

Fast track and ultrafast track cardiac anaesthesia appear to demonstrate improved outcomes without compromising patient safety. Their benefits include shorter intensive care unit stays, reduced duration of mechanical ventilation and lower health care costs. Regional anesthesia has played an important role in enhanced recovery pathways for other surgical services and allows for reduced systemic opioid use during intraoperative and postoperative care.

The anteromedial chest wall (i.e., the sternum and parasternal region) is innervated by the anterior branches of the intercostal nerves. These terminal anterior branches ascend in the parasternal region through the intercostal and pectoralis major muscles to innervate the superficial tissues. They can thus be targeted in one of two fascial planes: either deep into intercostal muscles and superficial to transversus thoracis muscles or superficial to the intercostal muscles and deep into pectoralis major muscle.

The sensory innervation of the thorax is provided by the 2nd through 6th intercostal nerves. The intercostal nerves terminate in anterior cutaneous branches, which divide into medial and lateral branches, providing innervation to the anterior chest wall. A pecto - intercostal nerve block targets the anterior intercostal nerves just lateral to the sternum in the interfascial plane between pectoralis major muscle and external intercostal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged more than 40 years old.
* scheduled for elective open-heart surgery including CABG with on pump cardiopulmonary bypass.

Exclusion Criteria:

* Patients with severe pulmonary hypertension and / or heart failure.
* Emergency or combined cardiac surgery.
* Patients with preoperative use of intra-aortic balloon pump.
* Patients with poor ventricular function less than 45 %.
* Patients with preoperative uncontrolled arrhythmia.
* Patients with moderate to severe hepatic and / or renal dysfunction.
* Patients with anticipated difficult airway.
* Severe obstructive and / or restrictive pulmonary function test.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
extubation time | up to 7 days postoperative
  duration of mechanical ventilation from the end of anaesthesia till fulfillment weaning criteria and extubated

SECONDARY OUTCOMES:
Postoperative mean arterial blood pressure measurement | within 24 hours postoperative
  mean arterial blood pressure measurement in mm Hg
Postoperative heart rate measurement | within 24 hours postoperative
  heart rate measurement in beat/min
ICU stay duration | up to 7 days postoperative
  from admission of ICU to discharge to ward
Postoperative pain measurement by numerical rating scale | within 24 hours postoperative
  Numerical Rating Scale for pain that ranged from (0 = no pain) to (10 = intolerable pain). If score is >3 will need analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Tarek Abdel Hay, Tanta, El Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No